CLINICAL TRIAL: NCT04697264
Title: Adipocytokines and Their Relationship to Obesity and Endometrial Cancer
Brief Title: Adipocytokines in Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: University of Surrey (Other)
Collaborators: Royal Surrey County Hospital NHS Foundation Trust (Other); GRACE Group (Other)
Responsible Party: Sponsor
Other Study IDs: SPON/2020/012/FHMS
Record Dates: First submitted 2020-12-01; First posted 2021-01-06 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Endometrial Cancer; Obesity
Keywords: Endometrial cancer; Obesity; Adiponectin; Leptin; TNF α; IL-6; IGF 1; IGF 2
MeSH Terms: conditions — Endometrial Neoplasms; Obesity | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and tissue (endometrial and adipose)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study - Patients with endometrial cancer: Potential participants will be identified in the Royal Surrey NHS Foundation trust - either seen here or referred here and receiving her treatment here for diagnosed endometrial cancer.
  Patients diagnosed with endometrial cancer will be identified through the Gynaecological Oncology Multi-Disciplinary Team meeting or by the Gynaecological Oncology or Medical Oncology teams.
  Blood sample will be collected on the day of the surgery when they are in the theatres and then repeated on day 1 post-operative in gynaecology ward and at 3/6 months post-surgery follow-up in clinic.
  For the women undergoing chemotherapy, blood sample will be procured prior to commencing chemotherapy and after 3rd (with the blood test before the fourth cycle of chemotherapy) and 6th cycles of chemotherapy.
  Interventions: Diagnostic Test: Blood and tissue sample collection from patients
- Control - patients without endometrial cancer, with benign gynaecological issues: Female patients being referred to Royal Surrey NHS foundation Trust for benign conditions (specifically not endometrial cancer) will be invited to participate as the control population.
  Interventions: Diagnostic Test: Blood and tissue sample collection from patients

INTERVENTIONS:
Diagnostic Test: Blood and tissue sample collection from patients — Blood and tissue sample (endometrial and adipose tissue) collection from endometrial cancer patients. Blood from all control patients, endometrial sample from benign patients having surgery for benign gynaecological conditions.

SUMMARY:
The number of women diagnosed with uterine cancer continues to rise each year. Since the early 1990s, there has been almost 55% rise in the United Kingdom (UK). 34% of endometrial cancer can be attributed to obesity. In the obese state, the function of adipose tissue deteriorates resulting in a state of chronic inflammation. Adipocytokine-related signalling pathways promote cancer development by causing inflammation, cell proliferation, DNA damage and by inhibiting apoptosis. The investigators postulate that adipocytokines levels are significantly different in uterine cancer patients of different weight categories and different grade/stage/ type of tumour.

Any woman attending the hospital with endometrial cancer and receiving treatment here will be invited to participate in the study. Consent will be sought to obtain 30mls (2 1/2 tablespoons) of venous blood at the time of surgery, on day 1 post-surgery and 3/6 months post-surgery during routine follow-up to check biomarker (adiponectin, leptin, tumour necrosis factor alpha, interleukin-6, Insulin-like growth factors 1 and 2) levels to see if the markers can be used to assess response to treatment. The investigators will also get consent to collect tissue - adipose tissue (after surgery) and uterine cancer tissue and lymph nodes (after histo-pathological evaluation) to assess for biomarkers. The investigators will also obtain blood samples from patients undergoing chemotherapy for advanced stage endometrial. All tissues procured will be anonymised and analysed at the oncology laboratory, Leggett building, University of Surrey and later correlated with patients' medical data as well as with tumour grade, stage and type. The investigators will also use archival tissue blocks stored at the same laboratory for analysis (previously consented for use in research). These are anonymised tissue and there is no link to patients' data.

The aim would be to ultimately find immuno-stimulatory/ suppressive biomarkers in order to develop novel diagnostic/ prognostic tools.

DETAILED DESCRIPTION:
1. BACKGROUND

   Endometrial cancer is the most common malignancy of the female genital tract. It is the fourth most common cancer in the UK with around 9,500 new cases in 2017, current lifetime risk being 1 in 36 women. The number of women diagnosed with endometrial cancer continues to rise each year. Since the early 1990s, uterine cancer incidence rates have increased by almost three-fifths (55%) in the UK (2015-2017). The association between endometrial cancer and obesity is well documented. 7.5% of all cancers in women in UK are attributable to being overweight / obese (BMI ≥25 kg/m2). For endometrial cancer, this risk rises to 34%. A review of meta-analyses showed endometrial cancer risk is 16% higher per 5 kg- gained during adulthood, 29% higher per 10cm increase in hip circumference and 27% higher per 10cm increase in waist circumference. This higher endometrial cancer risk with raised BMI is present in both pre- and post-menopausal women. Moreover, patients who are obese tend to have a poorer outcome with more co-morbidities than their non-obese counterparts.

   In the overweight and obese state, the function of the adipose tissue deteriorates resulting in a state of chronic inflammation. In this inflammatory state, adipocytes and macrophages secrete several molecules, adipokines and inflammatory cytokines, which may promote tumour development and angiogenesis and stimulate adhesions and migration of cells.

   Most implicated adipocytokines in the tumorigenesis pathway are adiponectin, leptin, tumour necrosis factor-α (TNF-α), Interleukin-6 (IL-6) and Insulin-like growth factor 1 and 2 (IGF 1 and 2).

   Adipocytokine related signalling pathways are important in the development of an inflammatory microenvironment for tumours. This process is thought to increase the risk of endometrial cancer by inducing cell proliferation and preventing cell apoptosis. Adiponectin, the most abundant adipokine, has been suggested to have anti-angiogenic, anti-inflammatory, and anti-apoptotic properties. Raised leptin levels in obese state promotes inflammation by stimulating the production of IL-6, TNFα as well as IL-1 and IL-126. Leptin and adiponectin secretion are counter-regulated in vivo. A study by Luhn et. al. has shown adiponectin to have inverse relationship with the risk of endometrial cancer and leptin to have a direct correlation.

   Also, in an inflammatory environment, macrophages secrete potent proinflammatory cytokines such as TNF-α and IL-6, which are known to activate numerous transcription factors that regulate the expression of genes involved in immune responses, anti-apoptosis, angiogenesis, and metastasis. The mechanisms of tumorigenesis are thought to be involved are free-radical production that cause DNA damage and impaired DNA repair.

   Research have further suggested that systemic levels of insulin-like growth factor (IGF) is dysregulated in obesity either due to increased IGF production or by down-regulation of IGF binding protein (IGFBP) production. IGF 1 is a growth and proliferation promotor and has inhibitory effects on cell death and is a major contributor in many neoplastic transformations.

   The above biomarkers are physiologically interrelated and are likely to reflect a more restricted number of underlying biological pathways. Possibly, they work in a synergistic capacity to modulate the risk of developing endometrial cancer. If specific patterns of cytokine expression were found to be predictive of adverse outcome, then the specific receptors may be targeted as a therapeutic option for endometrial cancer11. No study so far has looked at all these markers together in the serum and tissue samples of the same endometrial cancer patients to give a more wholesome idea about their effect on tumour genesis, progression and outcome. Therefore, this study is designed to assess the prognostic significance of these six biomarkers in the blood and tissue of endometrial cancer patients and co-relating the levels with their BMI and tumour type, after adjusting for age, parity, smoking status, menopausal status, use of hormone replacement therapy (HRT)/ hormonal contraception, and prevalence of diabetes and hypertension.
2. RATIONALE

   Development of novel biomarkers for a variety of uses including diagnosis, treatment monitoring and prognostication is on the Cancer Reform Strategy agenda and actively encouraged by the National Cancer Research Institute and Medical Research Council.

   Understanding how adipocytokines influence endometrial cancer risk may help to elucidate biological mechanisms important for the observed obesity-endometrial cancer association.
3. THEORITICAL FRAMEWORK

   As the incidence of endometrial cancer continues to rise there is a health need for a better diagnostic and prognostic approach.

   Studying the different biomarker levels in blood and cancer tissue will enable us to look for new targets that may be useful in the treatment and prognostication of this cancer.

   Also, if the levels of these markers change significantly post-treatment, the investigators can investigate if it will be possible to use these markers to assess response to treatment as follow-up for risk of recurrence forms an important part of the treatment protocol.
4. RESEARCH QUESTIONS / OBJECTIVES:

   To assess the relationship between the endometrial cancer and blood and tissue biomarkers in patients referred for endometrial cancer management to Royal Surrey NHS Foundation trust and to correlate with obesity and tumour characteristics.
5. STUDY DESIGN and METHODS of DATA COLLECTION AND DATA ANALYSIS

   5.1. Study design

   All patients being referred to the Royal Surrey NHS Foundation trust with diagnosed uterine cancer will be given the research information leaflet.

   Initially, an invitation letter will be sent alongside the patients' clinic appointment letter to inform them of the study and give them time for preliminary consideration of the study.

   Patients will then be approached in the outpatients' clinics after the initial consultation by the clinician. They will be given a participant information leaflet detailing the study rationale, methodology and analysis. Patients who agree to participate in the study will be asked to sign a consent form after explanation.

   Demographic data will be collected at the same time to correlate various risk factors associated with the development of uterine cancer. This data will be collected by:
   * A short patient interview (10 minutes)
   * Patients' medical notes Data from the interview will be directly entered into an existing departmental database for Gynaecological oncology which is password protected and stored on NHS computers. A copy of the data proformas from the interview will be filed in a secure room within the University department to allow for source data verification.

   Participants will then have 30mls (2 ½ tablespoons) of venous blood taken on the day of the surgery.

   Tissue samples from the participants undergoing hysterectomy will be collected as follows: the PI will collect any fresh tissue (adipose tissue) directly from theatre before fixing as it is not needed for establishing diagnosis and the uterine cancer tissue and lymph node will be collected by the PI after histo-pathological examination from the histo-pathology department after the diagnosis is established. All tissue processing will adhere to Human Tissue Authority (HTA) guidelines and will be performed at the Oncology laboratory at Leggett building at University of Surrey.

   The participants will have a repeat blood test (30mls) on day 1 post-surgery and at their 3 or 6 months routine post-surgery follow up appointment.

   For those participants who are recommended chemotherapy, the investigators will also ask consent to collect demographic data at the time of consultation and baseline blood sample (30mls venous blood) before commencing chemotherapy and after 3rd and 6th chemotherapy cycles to assess any changes in the biomarkers that may correlate with progression or regression of disease.

   The investigators will also obtain archival tissue blocks (of uterine cancer patients consented from a previous study for use during an appropriate ethics committee approved research) to help increase the number of recruitments for this study. Their demographic data with identification log will be made available to the PI only to assess for correlation between their data and the tissue diagnosis during analysis.

   5.2. Sample analysis

   ELISA will be used to assay bio-marker levels in blood samples.

   For tissue analysis the investigators will set up a tissue microarray (TMA). This will allow more uniform staining of the sample for immunohistochemistry with no inter-specimen variation of the staining method. Each case will be reviewed, and the area of interest (tumour) will be marked on the slide and cores from the areas of interest will be used to create the microarray block. Sections can then be cut from the microarray block and slides prepared for immune staining. The advantage of using this method is that the samples are subjected to the same conditions while being stained and the same part of a tumour can be reliably stained for several markers. Tissue sections from the TMA will be used for immune-staining and the expression of the markers of interest will be scored. Clinical data which is available on the cases will then be correlated with the histological and immunohistochemical scores and statistical analysis will be carried out.

   5.3. Data analysis

   Standard statistical analytical tools will be used to analyse the data. Relation between different variables will be sought with odds ratio, confidence interval and significance with P value (<0.05 significant). The Mann-Whitney U test will be used to assess differential expression of immune markers between tissue types -blood and tumour tissue. Correlation with clinical characteristics will be determined using univariate log-rank and multivariable Cox proportional hazards adjusting for age, stage, grade and histology.
6. SAMPLE AND RECRUITMENT

Potential participants will be identified in the Royal Surrey NHS Foundation trust - either seen here or referred here and receiving her treatment here for diagnosed endometrial cancer.

6.1. Sample size

The investigators will aim to recruit 30-60 patients with diagnosed endometrial cancer in the study. This sample size will also include archived tissue sample (formerly consented and stored in Leggett building, University of Surrey, for use in future ethical research).

6.2. Recruitment

All patients seen or referred with endometrial cancer at the Royal Surrey Oncology Department will be invited to participate in the study.

Patients will not receive any payments for participation in the study. The investigators aim to obtain all information and samples at the time of routine visits.

6.2.1. Sample identification

Patients diagnosed with endometrial cancer will be identified through the Gynaecological Oncology Multi-Disciplinary Team meeting or by the Gynaecological Oncology or Medical Oncology teams.

6.2.2. Consent

Written consent will be obtained after the patient has received the participant information leaflet and had the opportunity to discuss and ask questions about the study. Enough time will be given for the purpose. Patients must all have capacity to consent. Consent will be undertaken by clinicians on the Gynaecological Oncology team. If necessary, a translator or language line can be used.

Consent will also be taken for use of samples (anonymised and stored in Leggett building, University of Surrey following all regulations by HTA) for use in future research.

ELIGIBILITY:
Inclusion Criteria:

1. Women diagnosed with endometrial cancer
2. Age 18 or above
3. Of sound mind so they can give informed consent
4. Historical tissue sample/ blocks from previous cases in the laboratory in the University of Surrey, also be used if appropriate consent is in place.

Exclusion Criteria:

1. Under 18yrs age
2. Unable to give consent /denies consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population: All patients being referred to the Royal Surrey NHS Foundation Trust with diagnosed uterine cancer will be given the research information leaflet and invited to participate as the study population of the research.
  Control population: Female patients being referred to Royal Surrey NHS foundation Trust for benign conditions (specifically not endometrial cancer) will be invited to participate as the control population.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Surrey NHS Foundation Trust, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All personal information will be anonymised so that researchers except the Principal Investigator (PI) will be blinded to this information. At all times, the NHS Code of Confidentiality will be followed. Only the PI will have access to the 'key' to the patient identifiers connecting the samples to the clinical data of the patients which will be stored in a secured encrypted database on a NHS computer.

REFERENCES:
- [Background] Cancer Research UK Uterine Cancer Statistics http://www.cancerresearchuk.org/health-professional/cancer-statistics/statistics-by-cancer-type/uterine-cancer/incidence#heading-One
- [Background] Brown KF, Rumgay H, Dunlop C, Ryan M, Quartly F, Cox A, Deas A, Elliss-Brookes L, Gavin A, Hounsome L, Huws D, Ormiston-Smith N, Shelton J, White C, Parkin DM. The fraction of cancer attributable to modifiable risk factors in England, Wales, Scotland, Northern Ireland, and the United Kingdom in 2015. Br J Cancer. 2018 Apr;118(8):1130-1141. doi: 10.1038/s41416-018-0029-6. Epub 2018 Mar 23. PMID 29567982
- [Background] Kyrgiou M, Kalliala I, Markozannes G, Gunter MJ, Paraskevaidis E, Gabra H, Martin-Hirsch P, Tsilidis KK. Adiposity and cancer at major anatomical sites: umbrella review of the literature. BMJ. 2017 Feb 28;356:j477. doi: 10.1136/bmj.j477. PMID 28246088
- [Background] Luhn P, Dallal CM, Weiss JM, Black A, Huang WY, Lacey JV Jr, Hayes RB, Stanczyk FZ, Wentzensen N, Brinton LA. Circulating adipokine levels and endometrial cancer risk in the prostate, lung, colorectal, and ovarian cancer screening trial. Cancer Epidemiol Biomarkers Prev. 2013 Jul;22(7):1304-12. doi: 10.1158/1055-9965.EPI-13-0258. Epub 2013 May 21. PMID 23696194
- [Background] Nieman KM, Kenny HA, Penicka CV, Ladanyi A, Buell-Gutbrod R, Zillhardt MR, Romero IL, Carey MS, Mills GB, Hotamisligil GS, Yamada SD, Peter ME, Gwin K, Lengyel E. Adipocytes promote ovarian cancer metastasis and provide energy for rapid tumor growth. Nat Med. 2011 Oct 30;17(11):1498-503. doi: 10.1038/nm.2492. PMID 22037646
- [Background] Carbone F, La Rocca C, Matarese G. Immunological functions of leptin and adiponectin. Biochimie. 2012 Oct;94(10):2082-8. doi: 10.1016/j.biochi.2012.05.018. Epub 2012 Jun 26. PMID 22750129
- [Background] Shacter E, Weitzman SA. Chronic inflammation and cancer. Oncology (Williston Park). 2002 Feb;16(2):217-26, 229; discussion 230-2. PMID 11866137
- [Background] Carlson MJ, Thiel KW, Yang S, Leslie KK. Catch it before it kills: progesterone, obesity, and the prevention of endometrial cancer. Discov Med. 2012 Sep;14(76):215-22. PMID 23021376
- [Background] Gunter MJ, Hoover DR, Yu H, Wassertheil-Smoller S, Manson JE, Li J, Harris TG, Rohan TE, Xue X, Ho GY, Einstein MH, Kaplan RC, Burk RD, Wylie-Rosett J, Pollak MN, Anderson G, Howard BV, Strickler HD. A prospective evaluation of insulin and insulin-like growth factor-I as risk factors for endometrial cancer. Cancer Epidemiol Biomarkers Prev. 2008 Apr;17(4):921-9. doi: 10.1158/1055-9965.EPI-07-2686. PMID 18398032
- [Background] Dossus L, Lukanova A, Rinaldi S, Allen N, Cust AE, Becker S, Tjonneland A, Hansen L, Overvad K, Chabbert-Buffet N, Mesrine S, Clavel-Chapelon F, Teucher B, Chang-Claude J, Boeing H, Drogan D, Trichopoulou A, Benetou V, Bamia C, Palli D, Agnoli C, Galasso R, Tumino R, Sacerdote C, Bueno-de-Mesquita HB, van Duijnhoven FJ, Peeters PH, Onland-Moret NC, Redondo ML, Travier N, Sanchez MJ, Altzibar JM, Chirlaque MD, Barricarte A, Lundin E, Khaw KT, Wareham N, Fedirko V, Romieu I, Romaguera D, Norat T, Riboli E, Kaaks R. Hormonal, metabolic, and inflammatory profiles and endometrial cancer risk within the EPIC cohort--a factor analysis. Am J Epidemiol. 2013 Apr 15;177(8):787-99. doi: 10.1093/aje/kws309. Epub 2013 Mar 13. PMID 23492765
- [Background] Wang T, Rohan TE, Gunter MJ, Xue X, Wactawski-Wende J, Rajpathak SN, Cushman M, Strickler HD, Kaplan RC, Wassertheil-Smoller S, Scherer PE, Ho GY. A prospective study of inflammation markers and endometrial cancer risk in postmenopausal hormone nonusers. Cancer Epidemiol Biomarkers Prev. 2011 May;20(5):971-7. doi: 10.1158/1055-9965.EPI-10-1222. Epub 2011 Mar 17. PMID 21415362

RESULTS

PARTICIPANT FLOW:
Groups:
- Study - Patients With Endometrial Cancer: Potential participants will be identified in the Royal Surrey NHS Foundation trust - either seen here or referred here and receiving her treatment here for diagnosed endometrial cancer.
  Patients diagnosed with endometrial cancer will be identified through the Gynaecological Oncology Multi-Disciplinary Team meeting or by the Gynaecological Oncology or Medical Oncology teams.
  Blood sample were collected on the day of the surgery when they are in the theatres and then repeated on day 1 post-operative in gynaecology ward and at 6 months post-surgery follow-up in clinic.
  Endometrial and adipose tissue samples collected at the time of surgery.
- Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues: Female patients being referred to Royal Surrey NHS foundation Trust for benign conditions (specifically not endometrial cancer) will be invited to participate as the control population.
  One-time blood sample from all control patients. Endometrial sample, if available and consented, from benign patients having surgery for benign gynaecological conditions.
Period: Overall Study
Arm/Group | Study - Patients With Endometrial Cancer | Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study - Patients With Endometrial Cancer: Potential participants will be identified in the Royal Surrey NHS Foundation trust - either seen here or referred here and receiving her treatment here for diagnosed endometrial cancer.
  Patients diagnosed with endometrial cancer will be identified through the Gynaecological Oncology Multi-Disciplinary Team meeting or by the Gynaecological Oncology or Medical Oncology teams.
  Blood sample will be collected on the day of the surgery when they are in the theatres and then repeated on day 1 post-operative in gynaecology ward and at 3/6 months post-surgery follow-up in clinic.
  Endometrial and adipose tissue collection at the time of surgery.
- Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues: Female patients being referred to Royal Surrey NHS foundation Trust for benign conditions (specifically not endometrial cancer) will be invited to participate as the control population.
  Blood from all control patients, endometrial sample from benign patients having surgery for benign gynaecological conditions.
- Total: Total of all reporting groups
Arm/Group | Study - Patients With Endometrial Cancer | Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Full Range); unit: years] | 65.7 [34 to 95] | 66.1 [36 to 90] | 65.9 [34 to 95]
Sex/Gender, Customized [Number; unit: Female participants]
  All participants were female | 50 | 50 | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  3 Ethnicities: Caucasian | 43 | 48 | 91
  3 Ethnicities: Asian | 6 | 1 | 7
  3 Ethnicities: Afro-caribbean | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 50 | 50 | 100
Basal Metabolic Index (BMI) [Mean (Full Range); unit: kg/m2] | 32.1 [18.6 to 54] | 26.6 [18.5 to 43] | 29.35 [18.5 to 54]

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Circulating Levels of These Markers and Demographic Characteristics.
Description: Correlation between circulating levels of these markers and demographic characteristics such as age, parity, smoking status, menopausal status, medication use, use of HRT or hormonal contraception, the prevalence of diabetes and hypertension, any prior significant medical history or history of cancer and family history of cancer.
Time Frame: Data collected at baseline
Population: HRT usage counted among menopausal women only.
Measure: Count of Participants; unit: Participants
Arm/Group | Study - Patients With Endometrial Cancer | Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues
Number analyzed (Participants) | 50 | 50
Participants
  Menopause: Yes | 39 | 42
  Menopause: No | 11 | 8
  Smoking: Yes | 15 | 17
  Smoking: No | 35 | 33
  Hormonal contraception: Yes | 30 | 32
  Hormonal contraception: No | 20 | 18
  HRT among menopausal women: number analyzed (Participants) | 39 | 42
  HRT among menopausal women: Yes | 10 | 20
  HRT among menopausal women: No | 29 | 22
  Diabetes: Yes | 13 | 3
  Diabetes: No | 37 | 47
  Hypertension: Yes | 22 | 20
  Hypertension: No | 28 | 30
  Past history of cancer: Yes | 6 | 14
  Past history of cancer: No | 44 | 36
  Family history of cancer: Yes | 22 | 28
  Family history of cancer: No | 28 | 22
Statistical Analysis 1: Comparison: Study - Patients With Endometrial Cancer; The influence of age on adiponectin levels was analysed by dividing the population into binary groups (<60 years and >/= 60 years) to facilitate comparison; Test type: Other — Univariate linear regression was initially performed, followed by multivariate regression using the significant associations from the univariate analysis; p = 0.026, Regression, Linear — Adjustments to the p-values for multiple comparison were performed using Benjamini and Hochberg approach on 'R' and represented in the text as adjusted p-value
Statistical Analysis 2: Comparison: Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues; The influence of age on adiponectin levels was analysed by dividing the population into binary groups (<60years and >/=60years) to facilitate comparison; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.496, Regression, Linear — Adjustments to the p-values for multiple comparisons were performed using Benjamini and Hochberg approach on 'R'
Statistical Analysis 3: Comparison: Study - Patients With Endometrial Cancer vs Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues; The influence of age on leptin levels was analysed by dividing the population into binary groups (<60years and >/=60years) to facilitate comparison; Test type: Other — [test comment as in outcome 1, analysis 1]; p > 0.05, Regression, Linear
Statistical Analysis 4: Comparison: Study - Patients With Endometrial Cancer; The influence of age on IGF1 and 2 levels were analysed by dividing the population into binary groups (<60years and >/=60years) to facilitate comparison; Test type: Other — [test comment as in outcome 1, analysis 1]; p > 0.05, Regression, Linear — Adjustments to the p-values for multiple comparisons were performed using Benjamini and Hochberg approach on 'R'
Statistical Analysis 5: Comparison: Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues; [analysis description as in outcome 1, analysis 4]; Test type: Other — Univariate linear regression was initially performed, followed by multivariate regression using the significant associations from the univariate analysis. Adjustments to the p-values for multiple comparisons were performed using Benjamini and Hochberg approach on 'R'; p > 0.05, Regression, Linear — Adjustments to the p-values for multiple comparisons were performed using Benjamini and Hochberg approach on 'R'
Statistical Analysis 6: Comparison: Study - Patients With Endometrial Cancer; The influence of menopausal status on levels of adiponectin, leptin, IGF1 and 2 were analysed by dividing the population into binary groups (pre-menopausal and menopausal) to facilitate comparison; Test type: Other — [test comment as in outcome 1, analysis 1]; p > 0.05, Regression, Linear — Adjustments to the p-values for multiple comparisons were performed using Benjamini and Hochberg approach on 'R'
Statistical Analysis 7: Comparison: Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues; The influence of menopausal status on levels of adiponectin was analysed by dividing the population into binary groups (pre-menopausal and menopausal) to facilitate comparison; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.014, Regression, Linear — Adjustments to the p-values for multiple comparisons were performed using Benjamini and Hochberg approach on 'R'
Statistical Analysis 8: Comparison: Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues; The influence of menopausal status on levels of leptin was analysed by dividing the population into binary groups (pre-menopausal and menopausal) to facilitate comparison; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.006, Regression, Linear — Adjustments to the p-values for multiple comparisons were performed using Benjamini and Hochberg approach on 'R'
Statistical Analysis 9: Comparison: Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues; The influence of menopausal status on levels of IGF1 and IGF2 were analysed by dividing the population into binary groups (pre-menopausal and menopausal) to facilitate comparison; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.019, Regression, Linear — Adjustments to the p-values for multiple comparisons were performed using Benjamini and Hochberg approach on 'R'

2. Primary Outcome: Correlation Between Circulating Levels of These Markers (Day 0) and Cancer Characteristics in the Study Population, Using Linear Regresion.
Description: Data on endometrial cancer histological characteristics, including grade, stage, histology, LVSI, MELF and MSI were collected from histology reports.
  Endometrial cancer grade is based on glandular organisation: Grade 1 (<5% non-glandular), Grade 2 (6-50%), and Grade 3 (>50% non-glandular). Staging reflects cancer spread, from localised to distant involvement. Type 1 (70-80%) is estrogen-related cancer usually endometrioid histology, while Type 2 (10-20%) arises from atrophic endometrium, of non-endometrioid histology. A lower grade and stage and type 1 histology is associated with better prognosis. LVSI, cancer in lymphatic/vascular spaces of the myometrium, is an independent risk factor for recurrence. MELF (microcystic, elongated, fragmented myometrial invasion) correlates with larger tumours, deeper invasion, and LVSI. MSI indicates DNA mismatch repair defects and is linked to advanced histological features, such as deep invasion and high-grade endometrial cancers.
Time Frame: Data collected at baseline (day 0)
Population: Study population - patients with endometrial cancer
Measure: Count of Participants; unit: Participants
Arm/Group | Study - Patients With Endometrial Cancer
Number analyzed (Participants) | 50
Participants
  Grade 1 | 23
  Grade 2 | 13
  Grade 3 | 14
  Stage Ia+Ib | 41
  Stage II+III | 9
  Type1 histology | 36
  Type 2 histology | 14
  LVSI present | 15
  LVSI absent | 35
  MELF present | 6
  MELF absent | 29
  MSI present | 10
  MSI absent | 32
Statistical Analysis 1: Comparison: Study - Patients With Endometrial Cancer; Effects of LVSI on adiponectin levels were assessed using multivariate linear regression, with binary categorisations (presence and absence of LVSI) to facilitate comparisons; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.033, Regression, Linear — Adjustments to the p-values for multiple comparison were performed using Benjamini and Hochberg approach on 'R'
Statistical Analysis 2: Comparison: Study - Patients With Endometrial Cancer; Effects of MELF on TNF levels were assessed using multivariate linear regression, with binary categorisations (presence and absence of MELF) to facilitate comparisons; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.015, Regression, Linear — Adjustments to the p-values for multiple comparisons were performed using Benjamini and Hochberg approach on 'R'
Statistical Analysis 3: Comparison: Study - Patients With Endometrial Cancer; Effects of tumour grade (Grade 1/2), stage (Stage 1/ >/=1), histology (type 1 and type 2), and MSI (presence or absence) on the biomarker levels (adiponectin, leptin, IGF 1 and 2, IL6 and TNF) were assessed using multivariate linear regression, with binary categorisations to facilitate comparisons; Test type: Other — [test comment as in outcome 1, analysis 1]; p > 0.05, Regression, Linear — Adjustments to the p-values for multiple comparisons were performed using Benjamini and Hochberg approach on 'R'

3. Primary Outcome: The Difference in Circulating Plasma Levels of Adiponectin Between Study and Control Patients
Description: Plasma levels of adiponectin will be measured by ELISA in both the study and the control populations, and the results compared using linear regression tests.
Time Frame: The levels of the markers between the two groups of patients were compared at baseline (day 0) and presented here.
Population: Only baseline (D0/prior to surgery) levels of the markers have been listed below for comparison of baseline levels in cancer and control populations
Measure: Mean (Full Range); unit: μg/mL
Arm/Group | Study - Patients With Endometrial Cancer | Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues
Number analyzed (Participants) | 50 | 50
μg/mL | 5.9 [0.8 to 27.2] | 11 [3.1 to 29.6]
Statistical Analysis 1: Comparison: Study - Patients With Endometrial Cancer vs Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues; To compare biomarker levels between study and control populations, a linear regression model was used, adjusting for BMI, diabetes, and parity, which are the unmatched factors between the study and control groups. This adjustment aimed to mitigate the confounding impact of these factors, considering their individual influence on the risk of endometrial cancer; Test type: Other; p < 0.0001, Regression, Linear — Adjustments to the p-values for multiple comparison were performed using the Benjamini and Hochberg approach in 'R'

4. Primary Outcome: The Difference in Circulating Plasma Levels of Leptin, IGF1 and IGF2 Between Study and Control Patients.
Description: Plasma levels of leptin, IGF1 and IGF2 will be measured by ELISA in both the study and the control populations, and the results compared using linear regression tests.
Time Frame: The levels of the markers between the two groups of patients were compared at baseline (day 0) and presented here.
Population: as for outcome 3
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Study - Patients With Endometrial Cancer | Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues
Number analyzed (Participants) | 50 | 50
ng/mL
  Leptin | 61.2 [14.2 to 222.7] | 41.9 [8.9 to 135.6]
  IGF1 | 5.8 [0.0008 to 19.8] | 7.8 [0.9 to 26]
  IGF2 | 17.3 [2.2 to 51.2] | 19.3 [4.2 to 54.7]
Statistical Analysis 1: Comparison: Study - Patients With Endometrial Cancer vs Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues; [analysis description as in outcome 3, analysis 1]; Test type: Other; p > 0.05, Regression, Linear — Adjustments to the p-values for multiple comparison were performed using the Benjamini and Hochberg approach in 'R'

5. Primary Outcome: The Difference in Circulating Plasma Levels of IL6 and TNFα Between Study and Control Patients.
Description: Plasma levels of IL6 and TNFα will be measured by ELISA in both the study and the control populations, and the results compared using linear regression tests.
Time Frame: The levels of the markers between the two groups of patients were compared at baseline (day 0) and presented here.
Population: as for outcome 3
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Study - Patients With Endometrial Cancer | Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues
Number analyzed (Participants) | 50 | 50
pg/mL
  IL6 | 17.3 [2.2 to 51.2] | 19.3 [4.2 to 54.7]
  TNF | 118.8 [0 to 3504] | 418.8 [0 to 5182]
Statistical Analysis 1: Comparison: Study - Patients With Endometrial Cancer vs Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues; [analysis description as in outcome 3, analysis 1]; Test type: Other; p < 0.05, Regression, Linear — Adjustments to the p-values for multiple comparison were performed using the Benjamini and Hochberg approach in 'R'

6. Primary Outcome: Correlation Between the Markers and Study Patients' Obesity Status
Description: Correlation between the markers and patients' obesity status using WHO BMI subgroups.
Time Frame: Levels of the markers were compared with BMI of the study patients at baseline i.e. Day 0
Measure: Mean (Full Range); unit: kg/m2
Arm/Group | Study - Patients With Endometrial Cancer
Number analyzed (Participants) | 50
kg/m2 | 32.1 [18.6 to 54]
Statistical Analysis 1: Comparison: Study - Patients With Endometrial Cancer; The impact of BMI on biomarker levels was assessed by categorising the population into two groups-normal weight and overweight/obese-for straightforward comparison. Here, we present the associations between adiponectin and the BMI of the study population at baseline; Test type: Other; p > 0.05, Regression, Linear — Univariate linear regression was initially performed, followed by multivariate regression using the significant associations from the univariate analysis. P value <0.05 was considered significant
Statistical Analysis 2: Comparison: Study - Patients With Endometrial Cancer; The impact of BMI on biomarker levels was assessed by categorising the population into two groups-normal weight and overweight/obese-for straightforward comparison. Here, we present the associations between leptin and the BMI of the study population at baseline; Test type: Other; p = 0.09, Regression, Linear — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Study - Patients With Endometrial Cancer; The impact of BMI on biomarker levels was assessed by categorising the population into two groups-normal weight and overweight/obese-for straightforward comparison. Here, we present the association between IL6, TNFα, IGF1, and IGF2 and the BMI of the study population at baseline; Test type: Other; p > 0.05, Regression, Linear — [p-value comment as in outcome 6, analysis 1]

7. Primary Outcome: Correlation Between the Markers and Control Patients' Obesity Status
Description: Correlation between the markers and patients' obesity status using WHO BMI subgroups.
Time Frame: BMI was measured at baseline only for the control population.
Measure: Mean (Full Range); unit: kg/m2
Arm/Group | Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues
Number analyzed (Participants) | 50
kg/m2 | 26.6 [18.5 to 43]
Statistical Analysis 1: Comparison: Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues; The impact of BMI on biomarker levels was assessed by categorising the population into two groups-normal weight and overweight/obese-for straightforward comparison. Here, we present the associations between adiponectin and the BMI of the control population at baseline; Test type: Other; p = 0.004, Regression, Linear — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues; The impact of BMI on biomarker levels was assessed by categorising the population into two groups-normal weight and overweight/obese-for straightforward comparison. Here, we present the associations between leptin and the BMI of the control population at baseline; Test type: Other; p = 0.0002, Regression, Linear — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues; The impact of BMI on biomarker levels was assessed by categorising the population into two groups-normal weight and overweight/obese-for straightforward comparison. Here, we present the associations between IL6, TNFα, IGF1, and IGF2 and the BMI of the control population at baseline; Test type: Other; p > 0.05, Regression, Linear — [p-value comment as in outcome 6, analysis 1]

8. Secondary Outcome: Changes in Adiponectin Levels Before (Day 0) and After Surgery in the Study Population (at 6 Months).
Description: Levels of biomarkers were assessed at baseline, at day 1, and at 6 months post-surgery in endometrial cancer patients (study population). To assess the effect of treatment i.e. surgery +/- adjuvant treatment on the levels of the biomarkers, associations were sought between the levels of biomarkers before surgery (day 0) and 6 months post-surgery and the results have been presented here.
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: μg/mL
Groups:
- Study Population - at Baseline, Prior to Surgery: Blood sample were collected on the day of the surgery when they are in the theatres (day 0)
- Study Population - 6 Months Post Surgery: Study population was followed up 6 months post surgery and levels of the markers were analysed in their blood.
Arm/Group | Study Population - at Baseline, Prior to Surgery | Study Population - 6 Months Post Surgery
Number analyzed (Participants) | 50 | 50
μg/mL | 2.59 (0.086) | 2.26 (0.085)
Statistical Analysis 1: Comparison: Study Population - at Baseline, Prior to Surgery vs Study Population - 6 Months Post Surgery; Test type: Other; p = 0.0007, Mixed Models Analysis — Adjustments to the p-values for multiple comparisons were performed using Benjamini and Hochberg approach on 'R'

9. Secondary Outcome: Changes in Leptin, IGF1 and IGF2 Levels Before (Day 0) and After Surgery in the Study Population (at 6 Months).
Description: as for outcome 8
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Groups:
- Study Population - at Baseline, Prior to Suegry: Blood sample were collected on the day of the surgery when they are in the theatres (day 0)
Arm/Group | Study Population - at Baseline, Prior to Suegry | Study Population - 6 Months Post Surgery
Number analyzed (Participants) | 50 | 50
ng/mL
  Leptin | 5.42 (0.117) | 5.51 (0.115)
  IGF1 | 2.59 (0.113) | 2.94 (0.112)
  IGF2 | 3.93 (0.133) | 4.85 (0.132)
Statistical Analysis 1: Comparison: Study Population - at Baseline, Prior to Suegry vs Study Population - 6 Months Post Surgery; Leptin levels were compared between the day 0 and 6 months post-operative bloods; Test type: Other; p > 0.05, Mixed Models Analysis — Adjustments to the p-values for multiple comparisons were performed using Benjamini and Hochberg approach on 'R'
Statistical Analysis 2: Comparison: Study Population - at Baseline, Prior to Suegry vs Study Population - 6 Months Post Surgery; IGF1 levels were compared between the day 0 and 6 months post-operative bloods; Test type: Other; p = 0.004, Mixed Models Analysis — Adjustments to the p-values for multiple comparisons were performed using Benjamini and Hochberg approach on 'R'
Statistical Analysis 3: Comparison: Study Population - at Baseline, Prior to Suegry vs Study Population - 6 Months Post Surgery; IGF2 levels were compared between the day 0 and 6 months post-operative bloods; Test type: Other; p < 0.0001, Mixed Models Analysis — Adjustments to the p-values for multiple comparisons were performed using Benjamini and Hochberg approach on 'R'

10. Secondary Outcome: Changes in IL6 and TNFα Levels Before (Day 0) and After Surgery in the Study Population (at 6 Months).
Description: as for outcome 8
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Study Population - at Baseline, Prior to Suegry | Study Population - 6 Months Post Surgery
Number analyzed (Participants) | 50 | 50
pg/mL
  IL6 | 2.84 (0.419) | 3.01 (0.415)
  TNF | 3.70 (0.413) | 3.62 (0.409)

11. Secondary Outcome: Expression of These Biomarkers and Their Receptors in Endometrial Cancer Tissue and Adipose Tissue
Description: Expression of adiponectin, leptin, and their receptors were studied in endometrial cancer tissue and fat tissue using qRT-PCR. Fresh endometrial tissue was collected from 39 endometrial cancer and 5 control patients. Fresh adipose tissue was collected from these 39 endometrial cancer patients. Normal endometrium was used as a reference (calibrator sample) and the expressions of the biomarkers were calculated as fold changes compared to the expression in the calibrator sample using the delta-delta Ct formula. A higher fold change indicates greater expression of the marker in the study sample compared to the benign calibrator sample. This allowed for a standardised comparison of biomarker expression across different tissues, such as cancerous and adipose tissues.
Time Frame: The expression of these markers were investigated in the two tissue samples at baseline only (day 0).
Measure: Mean (Full Range); unit: fold change
Groups:
- Study Population - Endometrial Cancer Tissue: Fresh endometrial cancer tissue was collected for evaluation from 39 of the 50 endometrial cancer patients
- Study Population - Adipose Tissue: Fresh adipose tissue was collected from the same 39 patients from whom fresh endometrial samples was collected
Arm/Group | Study Population - Endometrial Cancer Tissue | Study Population - Adipose Tissue
Number analyzed (Participants) | 39 | 39
fold change
  Adiponectin / AdipoQ | 116.6 [0 to 2846.6] | 10165.2 [47.5 to 50360.3]
  AdipoQ receptor / ADIPOR1 | 3.15 [0 to 54.4] | 0.839 [0 to 6.34]
  AdipoQ receptor/ ADIPOR2 | 1.689 [0 to 20.8] | 1.741 [0 to 4.3]
  Leptin / Ob | 263.7 [0 to 4560.6] | 3765.1 [4.3 to 38967.9]
  Leptin receptor/ ObR | 0.328 [0 to 4.4] | 1.432 [0 to 6.43]
Statistical Analysis 1: Comparison: Study Population - Endometrial Cancer Tissue vs Study Population - Adipose Tissue; Expression of adiponectin was studied in endometrial cancer tissue and fat tissue using qRT-PCR; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Study Population - Endometrial Cancer Tissue vs Study Population - Adipose Tissue; Expression of leptin and their receptors were studied in endometrial cancer tissue and fat tissue using qRT-PCR; Test type: Other; p < 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: Study Population - Endometrial Cancer Tissue vs Study Population - Adipose Tissue; Expression of adiponectin receptors were studied in endometrial cancer tissue and fat tissue using qRT-PCR; Test type: Other; p > 0.05, t-test, 2 sided

12. Secondary Outcome: Expression of These Biomarkers and Their Receptors in Endometrial Cancer Tissue and Lymph Nodal Tissue
Description: The expression of adiponectin and leptin and their receptors were studied in endometrial cancer tissue and lymph node tissue using qRT-PCR. 12 FFPE lymph nodal tissue blocks were collected from patients with lymph node dissection. Fresh endometrial tissue was collected from 39 endometrial cancer and 5 control patients, however, the data for the 12 patients with lymph node dissection is presented here. Normal endometrium was used as a reference (calibrator sample) and the expressions of the biomarkers were calculated as fold changes compared to the expression in the calibrator sample using the delta-delta Ct formula. A higher fold change indicates greater expression of the marker in the study sample compared to the benign calibrator sample. This allowed for a standardised comparison of biomarker expression across different tissues, such as cancerous and lymph nodal tissue.
Time Frame: The expression of these markers were investigated in the two tissue samples at baseline only (day 0).
Measure: Mean (Full Range); unit: fold change
Groups:
- Study Population - Endometrial Cancer Tissue: Fresh endometrial cancer tissue was collected for evaluation from 39 of the 50 endometrial cancer patients. However, the data for the 12 patients with lymph node dissection is presented here.
- Study Population - Lymph Nodal Tissue: 12 FFPE lymph nodal tissue blocks were collected from patients with lymph node dissection.
Arm/Group | Study Population - Endometrial Cancer Tissue | Study Population - Lymph Nodal Tissue
Number analyzed (Participants) | 12 | 12
fold change
  Adiponectin / AdipoQ | 19.18 [0 to 102.2] | 653.235 [39.95 to 4803.93]
  ADIPOR1 | 0.69 [0 to 2.70] | 1.37 [0.08 to 13.59]
  ADIPOR2 | 1.35 [0 to 4.44] | 10.10 [0.61 to 94.03]
  Leptin / Ob | 97.57 [0 to 935.8] | 11448.21 [174.25 to 82094.62]
  Leptin receptor/ ObR | 0.15 [0 to 0.67] | 3.47 [0.28 to 34.3]
  IGF1 | 1.42 [0 to 9.2] | 4.5125 [0.04 to 51.63]
  IGF1R | 1.15 [0.13 to 3.74] | 7.49 [0.15 to 73.26]
  IGF2 | 8.20 [0 to 37] | 5.33 [0.06 to 61.82]
  IGF2R | 1.67 [0 to 3.15] | 0.73 [0.31 to 1.29]
  IL6 | 461.5 [0.3 to 4269.9] | 4100.21 [3.29 to 32881.76]
  IL6R | 4.56 [0.26 to 13.25] | 1238.38 [3.2 to 14263.1]
  TNF | 12.25 [0 to 85] | 23.46 [2.57 to 103.97]
  TNFR1A | 4.80 [0.37 to 10.36] | 144.9691667 [0.3 to 1332.57]
  TNFR1B | 6.11 [0.58 to 41.83] | 11.5525 [2.73 to 59.1]
Statistical Analysis 1: Comparison: Study Population - Endometrial Cancer Tissue vs Study Population - Lymph Nodal Tissue; Expression of adiponectin was studied in endometrial cancer tissue and lymph node tissue using qRT-PCR; Test type: Other; p = 0.0002, t-test, 2 sided
Statistical Analysis 2: Comparison: Study Population - Endometrial Cancer Tissue vs Study Population - Lymph Nodal Tissue; Expression of leptin was studied in endometrial cancer tissue and lymphnode tissue using qRT-PCR; Test type: Other; p = 0.011, t-test, 2 sided
Statistical Analysis 3: Comparison: Study Population - Endometrial Cancer Tissue vs Study Population - Lymph Nodal Tissue; The expression of IL6 receptor (IL6R) was studied in endometrial cancer tissue and lymphnode tissue using qRT-PCR; Test type: Other; p = 0.009, t-test, 2 sided
Statistical Analysis 4: Comparison: Study Population - Endometrial Cancer Tissue vs Study Population - Lymph Nodal Tissue; The expression of adiponectin receptor, leptin receptor, IGF1 and IGF 2 receptors, IL6, TNF, IGF1 and IGF2 were studied in endometrial cancer tissue and lymphnode tissue using qRT-PCR; Test type: Other; p > 0.05, t-test, 2 sided

13. Secondary Outcome: Correlation Between Circulating Adiponectin Levels and Their Expression in Endometrial Tissue.
Description: Correlation between circulating adiponectin levels (measured by ELISA) and their expression in endometrial tissue (measured by PCR). This was done for the 39 patients from whom we received the tissue sample.
Time Frame: At baseline, one time point measurement, Day 0
Measure: Mean (Full Range); unit: μg/ml
Groups:
- Circulating Levels of the Markers in Study Group ai.e.Patients With Endometrial Cancer: Blood sample were collected on the day of the surgery (day 0) and correlated with tissue levels
Arm/Group | Circulating Levels of the Markers in Study Group ai.e.Patients With Endometrial Cancer
Number analyzed (Participants) | 39
μg/ml | 5.76 [0.78 to 21.02]
Statistical Analysis 1: Comparison: Circulating Levels of the Markers in Study Group ai.e.Patients With Endometrial Cancer; Circulating adiponectin levels and the expression of these markers and their receptors in endometrial tissue were compared using correlation studies; Test type: Other; p > 0.05, Pearson's correlation test

14. Secondary Outcome: Correlation Between Circulating Leptin, IGF1 and IGF2 Levels and Their Expression in Endometrial Tissue.
Description: Correlation between circulating leptin, IGF1 and IGF2 levels (measured by ELISA) and their expression in endometrial tissue (measured by PCR). This was done for the 39 patients from whom we received the tissue sample.
Time Frame: At baseline, one time point measurement, Day 0
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Circulating Levels of the Markers in Study Group ai.e.Patients With Endometrial Cancer
Number analyzed (Participants) | 39
ng/mL
  Leptin | 57.99 [14.23 to 138.68]
  IGF1 | 5.73 [0.008 to 19.81]
  IGF2 | 16.35 [2.19 to 51.19]
Statistical Analysis 1: Comparison: Circulating Levels of the Markers in Study Group ai.e.Patients With Endometrial Cancer; Circulating leptin, IGF1 and IGF2 levels and the expression of these markers and their receptors in endometrial tissue were compared using Pearson's correlation studies; Test type: Other; p > 0.05, Pearson's correlation test

15. Secondary Outcome: Correlation Between Circulating IL6 and TNF Levels and Their Expression in Endometrial Tissue.
Description: Correlation between circulating IL6 and TNF levels (measured by ELISA) and their expression in endometrial tissue (measured by PCR). This was done for the 39 patients from whom we received the tissue sample.
Time Frame: At baseline, one time point measurement, Day 0
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Circulating Levels of the Markers in Study Group ai.e.Patients With Endometrial Cancer
Number analyzed (Participants) | 39
pg/mL
  IL6 | 31.71 [0 to 288.39]
  TNF | 57.13 [0 to 812.58]
Statistical Analysis 1: Comparison: Circulating Levels of the Markers in Study Group ai.e.Patients With Endometrial Cancer; Circulating IL6 and TNF levels and the expression of these markers and their receptors in endometrial tissue were compared using Pearson's correlation studies; Test type: Other; p > 0.05, Pearson's correlation test

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 6 months. Study patients were followed up at 6 months, control patients did not have any planned follow-up within the remits of the study.
Description: No adverse and / or serious events were reported as a direct outcome of the study.
Arm/Group | Study - Patients With Endometrial Cancer | Control - Patients Without Endometrial Cancer, With Benign Gynaecological Issues
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
1. Small sample size
2. The BMI of the study and the control samples were not matched
3. Control population not healthy population. Benign gynaecological conditions could influence their inflammatory marker levels, particularly in cases with endometrial issues such as abnormal uterine bleeding or endometrial hyperplasia.
4. Lack of multi-ethnicity in populations as >90% white population.
5. Same calibrator benign endometrial sample was used as calibrator sample for all three tissue types

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT04697264/Prot_SAP_000.pdf